CLINICAL TRIAL: NCT05874609
Title: Teaching Neuraxial Ultrasonography With a Virtual Reality Simulator of Spine: a Randomized Controlled Trial
Brief Title: Teaching Neuraxial Ultrasonography With a Virtual Reality Simulator of Spine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Clinical Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VR teaching
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Neuraxial Ultrasonography
Keywords: ultrasound-guided; neuraxial anesthesia; virtual reality
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): In the VR group, the participants spent 30 minutes with the VR spine simulator after receiving the didactic teaching session.
  Interventions: Other: Teaching with VR spine simulator
- Control group (Active Comparator): In the control group, the participants received a 30-min traditional didactic teaching session of spine ultrasonography.
  Interventions: Other: Traditional didactic teaching

INTERVENTIONS:
Other: Teaching with VR spine simulator — The participants spent 30 minutes with the VR spine simulator after receiving the didactic teaching session. The learning objective with the VR simulator is to review the 3D lumbar spine anatomic model，learn the sonoanatomy presented by a dynamic ultrasound scan of the sagittal and transverse plane, and practice a preprocedural ultrasound scan.
  Arms: VR group
Other: Traditional didactic teaching — A 30-min traditional didactic teaching session of spine ultrasonography. This session was consisted of general spine anatomy, sonographic technique and sonoanatomy, description of five key spine ultrasonographic views (transverse spinous process view, transverse interlaminar view, parasagittal oblique interlaminar view, parasagittal articular process view, parasagittal transverse process view), and a stepwise technique of preprocedural lumbar spine scan
  Arms: Control group

SUMMARY:
As one of the most extensively practiced regional block, neuraxial anesthesia is the basic skill for anesthesiologist to acquire. Recently, virtual reality (VR) has been proposed as a new simulation training method to enhance medical education. The aim of our study is to evaluate the practical skills of ultrasound scan and the satisfaction of students who undergo training using VR versus traditional didactic lecture.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized control trial to evaluate the performance of spine ultrasound scan after different training methods. Participants were randomly divided into two groups receiving different training methods: VR spine simulator or traditional didactic teaching. After the training, participants were required to perform a preprocedural spine ultrasound scan on healthy volunteers using the stepwise technique taught in the didactic teaching session. The participants needed to acquire three key ultrasound views during the scan and recognize the anatomic structures in three ultrasound views.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia residents in our department

Exclusion Criteria:

* having previous experience of spine ultrasonography training
* having previous experience of spine ultrasound scan.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite learning score | Up to 12 hours after ultrasound scan is finished
  Evaluating the self-assessed theoretical knowledge (10 points), self-assessed practical skills (20 points), self-assessed satisfaction (10 points) and willingness to applicate the technique in future practice (10 points).

SECONDARY OUTCOMES:
Time of scan | Up to 1 hour after ultrasound scan begins
  Defined as the time from the probe contacting the skin to acquiring the three key ultrasound views
Rate of anatomic structures recognition | Up to 12 hours after ultrasound scan is finished
  The correct rate of recognition among 12 anatomic structures (posterior complex, anterior complex, lamina and erector spinae in the parasagittal oblique interlaminar view, spinous process, lamina and erector spinae transverse spinous view, articular process, transverse process, posterior complex, anterior complex and spinal canal in the transverse interlaminar view)
Accuracy of depth measurement to the posterior complex | Up to 12 hours after ultrasound scan is finished
  The measurement was deemed correct if the error was less than 0.5cm